CLINICAL TRIAL: NCT06086353
Title: A Prospective, Single-arm, Multicenter, Observational Safety Surveillance Study of VyndaMx® (Tafamidis Capsule 61 mg) in Patients With Transthyretin Amyloid Cardiomyopathy (ATTR-CM) in India
Brief Title: A Study to Learn About Tafamidis in Patients With Transthyretin Amyloid Cardiomyopathy (ATTR-CM) in India
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B3461106; NCT06086353 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Transthyretin Amyloid Cardiomyopathy
Keywords: Safety surveillance; Tafamidis
MeSH Terms: interventions — tafamidis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with ATTR-CM in India
  Interventions: Drug: Tafamidis

INTERVENTIONS:
Drug: Tafamidis — Patients on tafamidis will be observed

SUMMARY:
The purpose of this study is to learn about the safety of Tafamidis for the treatment of Transthyretin amyloid cardiomyopathy (ATTR-CM) in India.

ATTR-CM is a condition that affects people's hearts. Transthyretin is a protein that is made in the liver. In some people this protein stops working and forms clumps called as amyloid. Transthyretin amyloid builds up in heart and stops the heart from pumping properly.

This study is seeking for participants who are:

* confirmed with ATTR-CM.
* given Tafamidis capsules to be taken by mouth.

The safety of Tafamidis capsules will be checked based on side effects. These side effects can happen within 6 months after taking Tafamidis. A side effect is something (expected or unexpected) that you feel was caused by a medicine or treatment you take. The study doctor will collect side effect information and put the information on patient's case form.

Follow-up of the patient's will be performed via clinic re-visit or over a call. It is not a rule for the participants to visit the clinic in this study.

This study will help to see if Tafamidis is safe.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥18 years) with diagnosis of cardiomyopathy of wild type or hereditary transthyretin-mediated amyloidosis (ATTR-CM).
* Patients to whom VyndaMx® Capsules is prescribed for the treatment of wild or hereditary ATTR-CM.

Exclusion Criteria:

* Patient with hypersensitivity to VyndaMx® Capsule or to any of the excipients in the product.
* Patients with rare hereditary problems of fructose intolerance.
* Patient who has a contraindication to VyndaMx® Capsules according to the approved local product label.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with ATTR-CM and prescribed with VyndaMx® Capsule 61 mg according to routine clinical practice at 3 centers in India and willing to participate will be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-06-06 (Actual)

PRIMARY OUTCOMES:
Number of Adverse events with Tafamidis | Baseline to 6 months
  The safety of VyndaMx® Capsules is the primary objective of the study and will be assessed based on Adverse events which would occur within 6 months from first dosing. Investigator will collect the safety related data until 6 months from first dosing of Tafamidis Capsules and will record these data on the Case report Form.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- India (3):
  - Sri Jayadeva Institute of Cardiovascular Sciences and Research, Bangalore, Karnataka
  - AIG Hospital, Hyderabad
  - Max Super Speciality Hospital, New Delhi

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B3461106